CLINICAL TRIAL: NCT07017491
Title: A Randomized, Open-Label, Cross-Over Study to Determine the Glycemic Index and Glycemic Load of Selected Melon Varieties in Healthy Adults
Brief Title: Determination of Glycemic Index and Glycemic Load of Selected Melon Varieties in Healthy Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rehman Medical Institute - RMI (Other)
Responsible Party: Principal Investigator, Naseer Ahmed, Associate Professor, Rehman Medical Institute - RMI
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GL/GI-NA_1V4
Record Dates: First submitted 2025-06-03; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-05

CONDITIONS: Glycemic Index; Glycemic Load
Keywords: GLYCEMIC LOAD

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single group (cross over) (Experimental): Participants will consume a glucose solution containing 50 grams of available carbohydrates. This will serve as the reference food to calculate the glycemic index (GI) of the test melons.
  Interventions: Other: Orange candy melon (Cucumis melo); Other: Rock melon ( Cucumis melo var.cantalupensis); Other: honey dew (cucumis melo L.)

INTERVENTIONS:
Other: Orange candy melon (Cucumis melo) — Participants will consume a portion of melon A containing 50g of available carbohydrates to evaluate postprandial glycemic response.
Other: Rock melon ( Cucumis melo var.cantalupensis) — Participants will consume a portion of melon B containing 50g of available carbohydrates to evaluate postprandial glycemic response.
Other: honey dew (cucumis melo L.) — Participants will consume a portion of melon C containing 50g of available carbohydrates to evaluate postprandial glycemic response.

SUMMARY:
This crossover study aims to determine and compare the glycemic index (GI) and glycemic load (GL) of different melon varieties in healthy adults. Using glucose as the reference food, participants will consume test portions of each melon variety containing equivalent amounts of available carbohydrates.

DETAILED DESCRIPTION:
This crossover study aims to determine and compare the glycemic index (GI) and glycemic load (GL) of different melon varieties in healthy adults. Using glucose as the reference food, participants will consume test portions of each melon variety containing equivalent amounts of available carbohydrates. Blood glucose levels will be monitored at regular intervals over a 2-hour period. The glycemic response will be used to calculate GI and GL values for each melon type. The study is intended to inform dietary recommendations for blood glucose management.

ELIGIBILITY:
Inclusion Criteria:

1) Healthy males and females aged 18-50 years. 2) Body mass index (BMI) :Normal BMI (18-24.9) 3) Willingness to follow dietary instructions and attend all testing sessions

* Exclusion Criteria:

  1. Individuals with known metabolic disorders (e.g., diabetes, metabolic syndrome).
  2. Use of medications or supplements affecting blood glucose.
  3. Allergy or intolerance to melon or glucose solutions.
  4. Not able to co ordinate

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Glycemic Index (GI) of Melon Varieties | 1 month
  The glycemic index of each melon variety will be calculated by comparing the incremental area under the blood glucose response curve (iAUC) over 2 hours after consumption of the test food, relative to glucose.

SECONDARY OUTCOMES:
Glycemic Load (GL) of Melon Varieties | 1 month
  Calculated using the formula:
  Glycemic Load = (Glycemic Index × amount of carbohydrate in a typical serving) ÷ 100

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.thenews.com.pk/print/899124-pakistan-ranks-3rd-in-prevalence-of-diabetes-in-world-after-china-and-india